CLINICAL TRIAL: NCT04497545
Title: The Influence of EMG-triggered Robotic Movement on Function and Mobility of Stroke
Brief Title: The Influence of EMG-triggered Robotic Movement on Function and Mobility of Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EGZOTech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Limanowa Trial
Record Dates: First submitted 2020-07-29; First posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Ischemic Stroke
Keywords: stroke,; rehabilitation,; EMG-triggered rehabilitation,; robotic-assisted movement,; gait
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): A four-week rehabilitation program (Monday to Friday) involving the hour of individual therapy and 30 minutes of therapy on the Luna EMG device.
  Interventions: Device: Luna EMG
- Control Group (Other): A four-week rehabilitation program (Monday to Friday) involving one hour of individual therapy and 30 minutes on lower limb rotor
  Interventions: Device: lower limb rotor

INTERVENTIONS:
Device: Luna EMG — The duration of the overall therapeutic intervention in both groups will be the same.
  Arms: Study Group
Device: lower limb rotor — The duration of the overall therapeutic intervention in both groups will be the same.
  Arms: Control Group

SUMMARY:
Rehabilitation of lower limbs after a stroke supported by robots aims to return to independence and minimize disability caused by the incident, but the results have been mixed. Objective of the study was to assess the changes in gait capabilities, muscle tone and daily activities in patients after a recent stroke who underwent a 6-week supervised rehabilitation process using exercises on the LUNA EMG neurorehabilitation robot. A total of 60 participants with impaired motor function and gait after subacute stroke were included in the study. Each patient was randomly assigned to an intervention (robot) or control group (RG or CG). All patients, except standard therapy, underwent 1 session of therapy per day, 5 days a week for 6 weeks. People with RG had 30 minutes of training sessions on the Luna EMG robot, while CG received exercises on the lower limb rotor. Patients were evaluated before the start of the study, and then after 2, 4 and 6 weeks of therapy using the Ashworth scale, Rivermead mobility index (RMI), Repty functional index, Time Up and Go test (TUG) and muscle circumference on the thigh.

ELIGIBILITY:
Inclusion Criteria:

* ischemic stroke,
* not later than 6 months ago,
* muscle strength of extensors and knee flexors on the Lovetta scale below 3,
* functional disorders of the lower limb,
* patient's condition allowing full understanding of commands
* continued/uninterrupted rehabilitation process for 28 days

Exclusion Criteria:

* cognitive impairment-lack of or poor cooperation between the patient and the therapist,
* stroke (more than 6 months after the incident),
* unstable clinical condition,
* muscle strength of knee extensors and flexors on the Lovett scale greater than or equal to 3,
* rigid fixed contractures within the lower limb,
* significant spasticity (Ashworth scale of 3 and above)

Ages: 29 Years to 91 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2019-02-24 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
Change in Timed up and go test results | baseline, after 4 weeks, after 6 weeks
  the test is performed from a sitting position. The patient on command is to get up from the chair to walk a distance of 3 meters, then turn back and sit on the chair
Change in Ashworth Scale results | baseline, after 4 weeks, after 6 weeks
  Measurement of resistance during passive knee flexion and extension
  Scorse range from 0 to 4, with 5 choices:
  Grade 0: No increase in muscle tone. Grade 1: Slight increase in muscle tone, manifested by a catch and release or by minimal.
  resistance when the affected part is moved in flexion or extension. Grade 2: More marked increase in muscle tone, but affected part(s) easily moved.
  Grade 3: Considerable increase in muscle tone, passive movement difficult. Grade 4: Affected part(s) rigid in flexion or extension. Higher values represent a worse outcome.
Change in Rivermeade Motor Assessment (RMA) | baseline, after 4 weeks, after 6 weeks
  The RMA assess functional mobility following stroke. Gross Function (RMA-Gf) : gait, balance, transfers.
  Each item is scored either yes "1" or no "0". It is based on Guttman scaling, which presumes that each subsequent item is of a more difficult nature. To advance to the next question, one must score (1) on an item, otherwise the test is stopped.
change in REPTY questionnair results | baseline, after 4 weeks, after 6 weeks
  a scoring scale for evaluation of ADL in hemiplegic patients. The higher score the more independent the patient is (the better)
Change in Tight Circumference | baseline, after 4 weeks, after 6 weeks
  thigh circumferences (5 and 15 centimeters above the patella),

CONTACTS AND LOCATIONS:
Locations (1):
- Rehstab, Limanowa, Malopolskie Voivodship, Poland

IPD SHARING:
Plan to Share IPD: Undecided